CLINICAL TRIAL: NCT01059721
Title: Treatment of Patella Dislocation in Childhood and Adolescence. Soft Tissue Realignment of the Tibial Insertion of the Patella Tendon. Long-term Outcome.
Brief Title: Outcome After Soft Tissue Realignment of the Tibial Insertion of the Patella Tendon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Frank Schneider, MD, consultant orthopedic surgeon, Medical University of Graz
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PatellaGraz
Record Dates: First submitted 2010-01-29; First posted 2010-02-01 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Patella Dislocation
Keywords: Centralisation; Patella dislocation; Open epiphyses; Malalignment syndrome; Relapse rate
MeSH Terms: conditions — Patellar Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Soft tissue realignment (Experimental): group cohort label
  Interventions: Procedure: Medialising insertion of patella tendon

INTERVENTIONS:
Procedure: Medialising insertion of patella tendon — surgical treatment of medialising tibial tuberosity

SUMMARY:
Soft tissue realignment of the tibial insertion of the patella tendon is a simple operative technique for treating dislocation of the patella in childhood and adolescence. It is performed in children with either recurrent dislocation or complicated primary dislocation in cases with malalignment or maltracking of the patella and a lateralised tibial tuberosity. It can be performed in patients with open epiphyses. We investigate long-term outcome after this procedure.

DETAILED DESCRIPTION:
Method. Investigation of the outcome of a relatively new method for centralisation of the insertion of the patella tendon in patients with open epiphyses. Using a soft tissue technique the patella tendon is released from the tibial tuberosity with the tendon still fixed to the distal periosteum. The tibial periosteum is split on the lateral border of the tibia distally. Together with lateral release this procedure releases the patella tendon which finds a new insertion more medially. Because the tendon is still fixed at the distal periosteum no additional fixation is needed and therefore no complications occur at the tibial apophysis due to osteosynthetic material. Full weight bearing is possible after 4 weeks and movement is not restricted.Results. From 1999 to 2004 a total of about 90 operations in about 80 patients for soft tissue centralisation of the distal insertion of the patella tendon were carried out on children and adolescents aged between 10 and 18 years old. This study is a retrospective analysis of the outcome after 6 to 10 years. Relevant outcome criteria will be evaluated with the occurrence of recurring dislocation, the Lysholm score, the Tegner activity scale and subjective measurement with the VAS scale and an additional functional outcome score, that we created especially for children. Eventual occurrence of growth disturbance or osteoarthritis will be documented be clinical or radiological features.

ELIGIBILITY:
Inclusion Criteria:

* Operative procedure soft tissue realignment performed between 1999 and 2004

Exclusion Criteria:

* Syndromal patella dislocation
* Genetic disorders

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Lyshom Score, Tegner-activity scale, VAS Pain assessment.Own examination form especially for children | 6 to 10 Years

SECONDARY OUTCOMES:
Radiological investigation | 6-10 years